CLINICAL TRIAL: NCT01790074
Title: MANUAL TREATMENT OF ACTIVE TRIGGER POINTS IN THE STERNOCLEIDOMASTOID MUSCLE IN PATIENTS WITH CERVICOGENIC HEADACHE: A PILOT RANDOMIZED CLINICAL TRIAL
Brief Title: Trigger Point Therapy in Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: César Fernández-de-las-Peñas (Other)
Collaborators: University of Alcala (Other)
Responsible Party: Sponsor-Investigator, César Fernández-de-las-Peñas, Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPA 2010
Record Dates: First submitted 2013-02-09; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Cervicogenic Headache
Keywords: cervicogenic headache; trigger point; sternocleidomastoid; manual therapy
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TrP therapy (Experimental): TrP manual therapy comprises different manual approaches, e.g., compression, stretching, or transverse friction massage applied over active TrPs in the sternocleidomastoid muscle
  Interventions: Other: TrP therapy
- TrP manual control therapy (Placebo Comparator): The treatment consisted of a simulation of the same TrP therapy treatment applied to the experimental group without the application of any therapeutic pressure.
  Interventions: Other: TrP manual control therapy

INTERVENTIONS:
Other: TrP therapy — TrP manual therapy comprises different manual approaches, e.g., compression, stretching, or transverse friction massage applied over active TrPs in the sternocleidomastoid muscle
  Arms: TrP therapy
Other: TrP manual control therapy — The treatment consisted of a simulation of the same TrP therapy treatment applied to the experimental group without the application of any therapeutic pressure.
  Arms: TrP manual control therapy

SUMMARY:
It is a pilot randomized controlled trial comparing real and simulated manual treatment of trigger points (TrPs) in patients with cervicogenic headache (CeH). The purpose of the current randomized clinical pilot trial was to determine the preliminary effects of TrP manual therapy in individuals with CeH with sternocleidomastoid muscle active TrPs as compared to manual contact over the muscle tissues.

DETAILED DESCRIPTION:
CeH pain has been mostly related to joint, disk and ligament pain from the upper cervical spine; however, clinicians should consider that the upper cervical spine also receives afferent inputs from muscles. In fact, the role of referred pain to the head elicited by muscle TrPs has received particular interest in recent years. No study has investigated the effectiveness of TrP manual therapy in patients with CeH exhibiting active TrPs. Investigators hypothesized that patients receiving a real TrP treatment will exhibit a greater reduction in pain, sensitivity, cervical range of motion and neck endurance than those receiving a manual control non-therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* unilateral pain starting in the neck and radiating to the frontal-temporal region
* pain aggravated by neck movement
* restricted cervical range of motion
* joint tenderness in at least one of the joints of the upper cervical spine (C1-C3)
* headache frequency of at least one per week over a period greater than 3 months
* active TrPs in the sternocleidomastoid muscle

Exclusion Criteria:

* other primary headaches (i.e., migraine, tension type-headache)
* bilateral headaches
* had received treatment for neck or head pain in the previous year
* presented any contraindications to manual therapy
* had pending legal action regarding their neck and head pain.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in headache intensity from baseline to one week after treatment | Baseline and one week after the intervention
  The intensity of head and neck pain was separately assessed with an 11-point numerical pain rate scale (NPRS, 0: no current pain, 10: maximum pain). It was recorded as a mean based on headaches experienced in the preceding week.

SECONDARY OUTCOMES:
Change in cervical range of motion from baseline to one week after treatment | Baseline and one week after the intervention
  Cervical range of motion was measured using a cervical range of motion (CROM) device. Subjects were asked to move their head as far as they could without pain in a stan¬dardized sequence: flexion, extension, affected/non-affected lateral flexion, and affected/non-affected rotation.
Change in pressure pain sensitivity from baseline to one week after treatment | Baseline and one week after the intervention
  Pressure pain thresholds (PPT), i.e., the amount of pressure where a sensation of pressure first changes to pain was assessed with an analogical algometer over C0-C1, C1-C2 and C2-C3 zygapophyseal joints on the symptomatic side.
Change in deep cervical flexors motor performance from baseline to one week after treatment | Baseline and one week after the intervention
  The motor performance of the deep cervical flexor muscles was tested in all patients by using the cervical flexor test (CCFT).

CONTACTS AND LOCATIONS:
Overall Officials: César Fernández-de-las-Peñas, PhD, DMSc, Study Chair — Universidad Rey Juan Carlos
Locations (1):
- University of Alcala, Alcalá de Henares, Madrid, Spain